CLINICAL TRIAL: NCT02483624
Title: A Single-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of 3,3'-Diindolylmethane (BR-DIM) in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: 3,3'-Diindolylmethane in Patients With Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06.02.107T
Record Dates: First submitted 2015-06-23; First posted 2015-06-29 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: SLE
MeSH Terms: interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Experimental): 10 patients 225 mg of BR-DIM. 2 capsules AM and 1 PM. 52 weeks duration.
  Interventions: Drug: BR-DIM
- High Dose (Experimental): 10 patients 375 mg of BR-DIM. 3 capsules AM and 2 PM. 52 weeks duration.
  Interventions: Drug: BR-DIM
- Placebo (Placebo Comparator): 10 patients receiving weight matched placebo. 5 for high dose and 5 for low dose. 52 weeks of weight matched pills.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BR-DIM — DIM, a condensation product of indole-3-carbinol (IC3), is a phytochemical that has activity against certain tumor cells. Observations in lupus-prone mice treated with indole-3-carbinol suggest that DIM might have favorable biologic and clinical effects in human SLE.
  Other Names: 3,3'-diindolylmethane
  Arms: High Dose; Low Dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a single center study of patients with inactive or mild SLE being performed to determine the safety, tolerability, and pharmacodynamics of DIM.

DETAILED DESCRIPTION:
This study is a single-blinded, placebo-controlled trial to determine the effects of DIM supplementation in patients with SLE. The DIM supplement to be used is BioResponse-DIM® (BR-DIM®), an absorption-enhanced formulation of proven bioavailability in animal testing and human trials. A total of 30 individuals will be enrolled into this 14-month study. Ten patients will be randomly assigned to the Low Dose Group [a daily dose of 225 mg of DIM from BR-DIM]. Ten patients will be randomly assigned to the High Dose Group [a daily dose of 375 mg of DIM from BR-DIM]. Ten patients will be randomly assigned to a matching placebo group, where 5 of these patients will receive matched placebo capsules equaling use in the Low Dose active group, and 5 will receive matched placebo equaling use in the High Dose active group. Each active capsule will deliver 75 mg of DIM from BR-DIM. Dosing will span 52 weeks. BR-DIM or comparably packaged placebo will be administered orally with meals twice per day. Placebo subjects randomized to the Low Dose group will take 2 placebo capsules in the am and 1 capsule in the pm and placebo subjects randomized to the high dose group will take 3 capsules in the am and 2 capsules in the pm. Low Dose active subjects will take 2 capsules in the am and 1 capsule in the pm. High Dose active subjects will take 3 capsules in the am and 2 capsules in the pm. Study subjects will be randomly assigned to one of the four treatment groups. Randomization procedures will be overseen by the staff of the North Shore Long Island Jewish General Clinical Research Center. The randomization schedule will be set up by the Bio-Statistics unit. The Investigator will contact the Research Pharmacy at North Shore University Hospital who will contact the Bio-Statistics unit once the subject signs the Informed Consent Form in order to learn which treatment regimen the subject is assigned to. Patients and control subjects will be given the appropriate amount of study medication at each visit to take home with them. Study personnel will monitor compliance by asking the patient to return any unused study medication at each visit for drug accountability. In addition, medication logs will be kept by the study subject and will be presented to the study coordinator at each visit. The subject, but not study personnel, will be blinded to the study drug assignments.

ELIGIBILITY:
Inclusion Criteria:

* Stable SLE disease activity for a period of at least 2 months prior to the Screening visit, based on the clinical judgment of the investigators
* History of measurable anti-dsDNA, anti-Sm, RNP, SS-A (anti-Ro), or SS-B (anti-La) autoantibodies
* Age > 18 and < 50
* Ability to understand the requirements of the study, provide written consent, and comply with the study protocol procedures
* A negative pregnancy test
* The use of contraception by fertile females
* A serum creatinine <1.8 mg/dL
* Serum hepatic transaminases < 1.25 times the upper limits of normal
* Hemoglobin > 9.5, WBC > 3.0, neutrophils > 1.2; platelets > 90,000

Exclusion Criteria:

* Immunosuppressive therapy (e.g. cyclophosphamide, cyclosporine, azathioprine, mycophenolate mofetil) or intravenous gamma globulin within 6 months of study entry
* Prior receipt of biologic agents, unless 9 months or 4 half-lives, whichever is greater, have passed since the last dose
* Prednisone > 10 mg/day (or its pharmacologic equivalent) within 2 months of randomization
* Pregnancy or the intent to conceive during the study or 3 months after study completion
* Concurrent medications such as danazol, DHEA, or other medications that affect estrogen levels or metabolism
* Nursing mothers
* Oral contraceptive use
* The presence of infection
* A history of poor procedural compliance
* Receipt of an investigational drug within 60 days of baseline
* Malignancy (except for basal cell carcinoma)
* Dose changes of steroids, anti-malarial drugs, or NSAID's within 4 weeks of randomization
* Peri- or post-menopausal state
* History of clinical evidence of active significant acute or chronic diseases (i.e., cardiovascular, pulmonary, untreated hypertension, anemia, gastrointestinal, hepatic, renal, neurological, cancer, or infectious diseases) that could confound the results of the study or put the subject at undue risk
* History of any other medical disease, laboratory abnormalities, or conditions that would make the subject (in the opinion of the investigators) unsuitable for the study
* Current drug or alcohol addiction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Routine clinical and laboratory parameters as well as SLE activity measurement with SELENA Systemic Lupus Erythematosus Disease Activity Index assessment. | 14 months
  Routine clinical and laboratory parameters as well as SLE activity measurement with SELENA Systemic Lupus Erythematosus Disease Activity Index assessment.
Estradiol Hydroxylation Pathways | 14 months
  Measure alterations in the ratio of 2-hydroxyestrone/ 16alpha-hydroxyestrone (2-OHE/16alpha-OHE) in the urine.
Autoantibody Production | 14 Months
  Routine lab testing to determine whether DIM supplementation will decrease autoantibody production
T and B Lymphocytes | 14 Months
  Qualitative and quantitative abnormalities in B- and T-lymphocytes abound in human SLE. In this aim, phenotypic analyses of B- and T-lymphocyte subsets as well as functional analyses will be ascertained in order to evaluate the effects of DIM on these parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Furie, MD, Principal Investigator — NorthShore-LIJ Health System

REFERENCES:
- [Background] Roubinian JR, Talal N, Greenspan JS, Goodman JR, Siiteri PK. Effect of castration and sex hormone treatment on survival, anti-nucleic acid antibodies, and glomerulonephritis in NZB/NZW F1 mice. J Exp Med. 1978 Jun 1;147(6):1568-83. doi: 10.1084/jem.147.6.1568. PMID 308087
- [Background] Roubinian J, Talal N, Siiteri PK, Sadakian JA. Sex hormone modulation of autoimmunity in NZB/NZW mice. Arthritis Rheum. 1979 Nov;22(11):1162-9. doi: 10.1002/art.1780221102. No abstract available. PMID 508370
- [Background] Carlsten H, Nilsson N, Jonsson R, Backman K, Holmdahl R, Tarkowski A. Estrogen accelerates immune complex glomerulonephritis but ameliorates T cell-mediated vasculitis and sialadenitis in autoimmune MRL lpr/lpr mice. Cell Immunol. 1992 Oct 1;144(1):190-202. doi: 10.1016/0008-8749(92)90236-i. PMID 1394437
- [Background] Petri M. Exogenous estrogen in systemic lupus erythematosus: oral contraceptives and hormone replacement therapy. Lupus. 2001;10(3):222-6. doi: 10.1191/096120301676707393. PMID 11315357
- [Background] Bradlow HL, Telang NT, Sepkovic DW, Osborne MP. 2-hydroxyestrone: the 'good' estrogen. J Endocrinol. 1996 Sep;150 Suppl:S259-65. PMID 8943806
- [Background] Swaneck GE, Fishman J. Covalent binding of the endogenous estrogen 16 alpha-hydroxyestrone to estradiol receptor in human breast cancer cells: characterization and intranuclear localization. Proc Natl Acad Sci U S A. 1988 Nov;85(21):7831-5. doi: 10.1073/pnas.85.21.7831. PMID 3186693
- [Background] Lahita RG, Bradlow HL, Kunkel HG, Fishman J. Increased 16 alpha-hydroxylation of estradiol in systemic lupus erythematosus. J Clin Endocrinol Metab. 1981 Jul;53(1):174-8. doi: 10.1210/jcem-53-1-174. PMID 7240374
- [Background] Michnovicz JJ, Bradlow HL. Altered estrogen metabolism and excretion in humans following consumption of indole-3-carbinol. Nutr Cancer. 1991;16(1):59-66. doi: 10.1080/01635589109514141. PMID 1656396
- [Background] Bradlow HL, Michnovicz J, Telang NT, Osborne MP. Effects of dietary indole-3-carbinol on estradiol metabolism and spontaneous mammary tumors in mice. Carcinogenesis. 1991 Sep;12(9):1571-4. doi: 10.1093/carcin/12.9.1571. PMID 1893517
- [Background] Michnovicz JJ, Adlercreutz H, Bradlow HL. Changes in levels of urinary estrogen metabolites after oral indole-3-carbinol treatment in humans. J Natl Cancer Inst. 1997 May 21;89(10):718-23. doi: 10.1093/jnci/89.10.718. PMID 9168187
- [Background] Chen DZ, Qi M, Auborn KJ, Carter TH. Indole-3-carbinol and diindolylmethane induce apoptosis of human cervical cancer cells and in murine HPV16-transgenic preneoplastic cervical epithelium. J Nutr. 2001 Dec;131(12):3294-302. doi: 10.1093/jn/131.12.3294. PMID 11739883
- [Background] Rosen CA, Woodson GE, Thompson JW, Hengesteg AP, Bradlow HL. Preliminary results of the use of indole-3-carbinol for recurrent respiratory papillomatosis. Otolaryngol Head Neck Surg. 1998 Jun;118(6):810-5. doi: 10.1016/S0194-5998(98)70274-8. PMID 9627242
- [Background] Bell MC, Crowley-Nowick P, Bradlow HL, Sepkovic DW, Schmidt-Grimminger D, Howell P, Mayeaux EJ, Tucker A, Turbat-Herrera EA, Mathis JM. Placebo-controlled trial of indole-3-carbinol in the treatment of CIN. Gynecol Oncol. 2000 Aug;78(2):123-9. doi: 10.1006/gyno.2000.5847. PMID 10926790
- [Background] Auborn KJ, Qi M, Yan XJ, Teichberg S, Chen D, Madaio MP, Chiorazzi N. Lifespan is prolonged in autoimmune-prone (NZB/NZW) F1 mice fed a diet supplemented with indole-3-carbinol. J Nutr. 2003 Nov;133(11):3610-3. doi: 10.1093/jn/133.11.3610. PMID 14608082
- [Background] Theofilopoulos AN, Dixon FJ. Murine models of systemic lupus erythematosus. Adv Immunol. 1985;37:269-390. doi: 10.1016/s0065-2776(08)60342-9. No abstract available. PMID 3890479
- [Background] Anderton MJ, Manson MM, Verschoyle R, Gescher A, Steward WP, Williams ML, Mager DE. Physiological modeling of formulated and crystalline 3,3'-diindolylmethane pharmacokinetics following oral administration in mice. Drug Metab Dispos. 2004 Jun;32(6):632-8. doi: 10.1124/dmd.32.6.632. PMID 15155555
- [Background] Reed GA, Sunega JM, Sullivan DK, Gray JC, Mayo MS, Crowell JA, Hurwitz A. Single-dose pharmacokinetics and tolerability of absorption-enhanced 3,3'-diindolylmethane in healthy subjects. Cancer Epidemiol Biomarkers Prev. 2008 Oct;17(10):2619-24. doi: 10.1158/1055-9965.EPI-08-0520. PMID 18843002